CLINICAL TRIAL: NCT00308516
Title: A Phase II Study of 5-Fluorouracil, Bevacizumab (Avastin), and Radiation in the Preoperative or Adjuvant Treatment of Patients With Stage II / III Rectal Cancer
Brief Title: 5-Fluorouracil, Bevacizumab, and Radiation Followed by Modified FOLFOX6 and Bevacizumab in Stage II/III Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 65; AVF3105s (Other: Genentech-Roche)
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Rectal Cancer; Cancer of the Rectum; Colorectal Cancer
Keywords: Rectal Cancer; Cancer of the Rectum; Colorectal Cancer; Bevacizumab
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Radiotherapy; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A - Preoperative (Experimental): Each patient enrolled in the preoperative cohort received 5-fluorouracil (5-FU) 225 mg/m2 as a continuous infusion (IVCI) on days 1-42 through a portable infusion pump and central venous catheter. Bevacizumab 5 mg/kg was administered intravenously (IV) on days 1 and 15. Additionally these patients received radiation therapy to 50.4 Gy (1.8 Gy/day or 28 fractions) Monday through Friday during weeks 1-6.
  At least 8 weeks after surgery, patients in cohort A began 4 months of chemotherapy and bevacizumab. This adjuvant treatment consisted of 5-FU 400 mg/m2 IV bolus over 2-4 minutes followed by 2400 mg/m2 IVCI over 46 hours, leucovorin 350 mg as a 2-hour infusion, oxaliplatin 85 mg/m2 IV (modified FOLFOX6) and bevacizumab 5 mg/kg IV all on days 1 and 15 of each cycle.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Procedure: Radiation Therapy; Drug: Oxaliplatin; Drug: Leucovorin
- Cohort B - Combined Modality (Experimental): All patients enrolled in cohort B received 5-fluorouracil (5-FU) 225 mg/m2 IVCI on days 1-42. Bevacizumab was administered at 5 mg/kg IV on day 1 every 2 weeks. These patients also received radiation to 50.4 Gy (1.8 Gy/day or 28 fractions)Monday through Friday during weeks 1-6.
  Six weeks after the completion of adjuvant 5-FU/radiation, patients began treatment with 5-FU 400 mg/m2 IV bolus over 2-4 minutes followed by 2400 mg/m2 IVCI over 46 hours, leucovorin 350 mg as a 2-hour infusion, oxaliplatin 85 mg/m2 IV (modified FOLFOX6) and bevacizumab 5 mg/kg IV all on days 1 and 15 of each cycle.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Procedure: Radiation Therapy; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: 5-Fluorouracil — Combined Modality Treatment:
  fluorouracil 225mg/m2 IV continuous infusion days 1-42
  Systemic Treatment:
  5-fluorouracil 400 mg/m2 bolus 5-fluorouracil 2400 mg/m2 over 46 hours days 1 and 15
  Other Names: Fluorouracil; Efudex; 5-FU
Drug: Bevacizumab — Combined Modality Treatment:
  bevacizumab 5mg/kg IV infusion days 1, 15, and 29
  Systemic Treatment:
  bevacizumab 5 mg/kg days 1 and 15
  Other Names: Avastin
Procedure: Radiation Therapy — radiation 1.8 Gy/day or 28 fractions weeks 1-6
Drug: Oxaliplatin — Systemic Treatment:
  oxaliplatin 85 mg/m2 days 1 and 15
  Other Names: Eloxatin
Drug: Leucovorin — Systemic Treatment:
  leucovorin 350 mg prior to FU on days 1 and 15
  Other Names: Folinic acid

SUMMARY:
This phase II trial will investigate the combination of adjuvant 5-fluorouracil, radiation, and bevacizumab in patients with stage II and III rectal cancer, followed by FOLFOX6 and bevacizumab. Fluorouracil (FU) has proven to be an effective and safe regimen in the treatment of stage II and III rectal cancer. Recent evidence has proven fluorouracil/leucovorin (FL) in combination with bevacizumab is superior to FL alone and when combined with irinotecan is superior to (irinotecan plus fluorouracil/leucovorin (IFL) alone. This trial will be one of the first clinical trials to evaluate a combination of targeted therapy, radiation, and chemotherapy in the adjuvant treatment of a common solid tumor.

DETAILED DESCRIPTION:
All eligible patients will receive combined modality treatment initially. Systemic treatment will begin 4-6 weeks after completion of the Combined Modality portion and will complete 4 cycles of a 4 week regimen. Patients with no evidence of disease following systemic therapy may continue single agent bevacizumab for up to one year. After all treatment is completed, patients will be re-evaluated with imaging to establish a new baseline. Patients will be re-evaluated thereafter for up to a total of 5 years.

Combined Modality Treatment:

* bevacizumab 5mg/kg IV infusion days 1, 15, and 29
* fluorouracil 225mg/m2 IV continuous infusion days 1-42
* radiation 1.8 Gy/day or 28 fractions weeks 1-6

Systemic Treatment:

* 5-fluorouracil 400 mg/m2 bolus
* 5-fluorouracil 2400 mg/m2 over 46 hours days 1 and 15
* leucovorin 350 mg prior to FU on days 1 and 15
* oxaliplatin 85 mg/m2 days 1 and 15
* bevacizumab 5 mg/kg days 1 and 15

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage I or II rectal cancer
* Patients must be candidates for preoperative or adjuvant chemoradiation.
* Patients enrolling in the adjuvant chemoradiation cohort must have undergone surgical resection of the primary rectal tumor between 28 and 56 days (i.e., 4-8 weeks) prior to study treatment.
* ECOG performance status 0-1
* Adequate bone marrow, liver, and kidney function
* At least 18 years of age
* Able to give written informed consent

Exclusion Criteria:

* Treatment with prior chemotherapy or radiation for rectal cancer
* History of myocardial infarction
* Uncontrolled hypertension, unstable angina, congestive heart failure, serious cardiac arrhythmia requiring medication or peripheral vascular disease
* History of stroke within 6 months
* History of abdominal fistula, gastrointestinal perforation, or intrabdominal abscess within 6 months
* Symptomatic sensory or peripheral neuropathy
* Prior treatment with anti-angiogenic agents
* Prior malignancy in the past 5 years
* Active infections or serious underlying medical condition
* Major surgery less than 28 days prior
* Women who are pregnant or lactating
* Thrombolytic therapy within 10 days of starting bevacizumab
* PEG tube, G-tube, or external biliary stents
* Proteinuria
* Non healing wound, ulcer or fracture
* History of bleeding diathesis or coagulopathy
* Hemoptysis
* Participation in another experimental trial within 28 days
* Uncontrolled anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (14):
- United States (14):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Background] Spigel DR, Bendell JC, McCleod M, Shipley DL, Arrowsmith E, Barnes EK, Infante JR, Burris HA 3rd, Greco FA, Hainsworth JD. Phase II study of bevacizumab and chemoradiation in the preoperative or adjuvant treatment of patients with stage II/III rectal cancer. Clin Colorectal Cancer. 2012 Mar;11(1):45-52. doi: 10.1016/j.clcc.2011.04.002. Epub 2011 Aug 15. PMID 21840771

RESULTS

PARTICIPANT FLOW:
Groups:
- Preoperative 5FU/Radiation/Bevacizumab: Each patient enrolled in the preoperative cohort received 5-fluorouracil (5-FU) 225 mg/m2 as a continuous infusion (IVCI) on days 1-42 through a portable infusion pump and central venous catheter. Bevacizumab 5 mg/kg was administered intravenously (IV) on days 1 and 15. Additionally these patients received radiation therapy to 50.4 Gy (1.8 Gy/day or 28 fractions) Monday through Friday during weeks 1-6.
  At least 8 weeks after surgery, patients in cohort A began 4 months of chemotherapy and bevacizumab. This adjuvant treatment consisted of 5-FU 400 mg/m2 IV bolus over 2-4 minutes followed by 2400 mg/m2 IVCI over 46 hours, leucovorin 350 mg as a 2-hour infusion, oxaliplatin 85 mg/m2 IV (modified FOLFOX6) and bevacizumab 5 mg/kg IV all on days 1 and 15 of each cycle.
- Postoperative 5FU/Radiation/Bevacizumab: All patients enrolled in cohort B received 5-fluorouracil (5-FU) 225 mg/m2 IVCI on days 1-42. Bevacizumab was administered at 5 mg/kg IV on day 1 every 2 weeks. These patients also received radiation to 50.4 Gy (1.8 Gy/day or 28 fractions)Monday through Friday during weeks 1-6.
  Six weeks after the completion of adjuvant 5-FU/radiation, patients began treatment with 5-FU 400 mg/m2 IV bolus over 2-4 minutes followed by 2400 mg/m2 IVCI over 46 hours, leucovorin 350 mg as a 2-hour infusion, oxaliplatin 85 mg/m2 IV (modified FOLFOX6) and bevacizumab 5 mg/kg IV all on days 1 and 15 of each cycle.
Period: Overall Study
Arm/Group | Preoperative 5FU/Radiation/Bevacizumab | Postoperative 5FU/Radiation/Bevacizumab
Started | 35 | 31
Completed | 6 | 10
Not Completed | 29 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative 5FU/Radiation/Bevacizumab | Postoperative 5FU/Radiation/Bevacizumab | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Median (Full Range); unit: years] | 57 [26 to 82] | 56 [31 to 76] | 57 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 26 | 15 | 41
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 66

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS), The Proportion of Patients Predicted to be Alive Without Evidence of Disease Recurrence 24 Months After Completion of Protocol Treatment
Description: The Proportion of Patients Predicted to be Alive Without Evidence of Disease Recurrence 24 Months After Completion of Protocol Treatment
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Preoperative 5FU/Radiation/Bevacizumab | Postoperative 5FU/Radiation/Bevacizumab
Number analyzed (Participants) | 35 | 31
percentage of participants | 85 [67 to 93] | 97 [79 to 100]

2. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Overall Survival (OS) is defined ad the Length of time, in months, that patients were alive from their first date of protocol treatment until death.
Time Frame: 24 months
Population: The median survival was not reached for either of the cohorts
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative 5FU/Radiation/Bevacizumab | Postoperative 5FU/Radiation/Bevacizumab
Number analyzed (Participants) | 35 | 31
months | NA [NA to NA] — The 95% CI is not estimable by Kaplan-Meier method since the median survival was not reached by the 24 month follow up period | NA [NA to NA] — The 95% CI is not estimable by Kaplan-Meier method since the median survival was not reached by the 24 month follow up period

ADVERSE EVENTS:
Arm/Group | Preoperative 5FU/Radiation/Bevacizumab | Postoperative 5FU/Radiation/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 18/35 | 15/31
Other Adverse Events (participants affected / at risk) | 35/35 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative 5FU/Radiation/Bevacizumab (N=35) | Postoperative 5FU/Radiation/Bevacizumab (N=31)
Infection - Pelvis (Infections and infestations) | 1 (1) | 0 (0)
Infection - NOS (Infections and infestations) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction - GI (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain - Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fistula, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perforation, GI (Gastrointestinal disorders) | 1 (1) | 2 (2)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain - Abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Vulvar excoriation
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection - GI (Infections and infestations) | 0 (0) | 2 (2)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection - Skin (Infections and infestations) | 1 (1) | 0 (0)
Mental Status (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Surgery/Intraoperative Injury - Prostate (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection - Postoperative (Infections and infestations) | 1 (1) | 0 (0)
Wound Complication (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection - Renal/Genitourinary (Infections and infestations) | 1 (1) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 (2) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative 5FU/Radiation/Bevacizumab (N=35) | Postoperative 5FU/Radiation/Bevacizumab (N=31)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2 (5) | 4 (5)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (8)
ALT (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Anorexia (Gastrointestinal disorders) | 15 (19) | 11 (24)
AST (Metabolism and nutrition disorders) | 4 (9) | 2 (3)
Bilirubin (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Rigor/Chills (General disorders) | 2 (2) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 9 (16) | 4 (6)
Cold Sensitivity (General disorders) | 2 (2) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (5)
Constipation (Gastrointestinal disorders) | 9 (21) | 8 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Dehydration (Gastrointestinal disorders) | 9 (10) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 24 (54) | 27 (70)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (13) | 4 (7)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (4)
Edema - Limb (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 29 (72) | 22 (66)
Fever (General disorders) | 3 (3) | 5 (7)
Rectal Drainage (Gastrointestinal disorders) | 2 (3) | 2 (2)
Hand-Foot (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (8)
Hemoglobin (Blood and lymphatic system disorders) | 22 (65) | 18 (47)
Hemorrhage - Hematuria (Renal and urinary disorders) | 2 (6) | 0 (0)
Hemorrhage - Gums (Blood and lymphatic system disorders) | 0 (0) | 2 (5)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 7 (17) | 6 (11)
Hemorrhage - GI (Gastrointestinal disorders) | 5 (6) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 2 (6) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (13) | 7 (29)
Hypertension (Cardiac disorders) | 6 (12) | 7 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (8) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 2 (4)
Infection - Postoperative (Infections and infestations) | 3 (3) | 0 (0)
Infection - GI (Infections and infestations) | 0 (0) | 3 (5)
Infection - Skin (Infections and infestations) | 3 (3) | 2 (2)
Infection - Upper Respiratory (Infections and infestations) | 3 (9) | 3 (4)
Infection - Renal/Genitourinary (Infections and infestations) | 7 (7) | 3 (3)
Infection with Normal ANC (Infections and infestations) | 2 (2) | 5 (5)
Insomnia (General disorders) | 4 (11) | 7 (10)
Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Leukocytes (Immune system disorders) | 22 (75) | 21 (72)
Mental Status (Psychiatric disorders) | 0 (0) | 2 (3)
Mood Alteration - Anxiety (Psychiatric disorders) | 5 (16) | 2 (2)
Mood Alteration - Depression (Psychiatric disorders) | 4 (15) | 2 (2)
Mucositis/Stomatitis (Gastrointestinal disorders) | 15 (19) | 12 (19)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (39) | 18 (38)
Neuropathy - Motor (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophils (Immune system disorders) | 14 (32) | 15 (36)
Pain - NOS (General disorders) | 25 (79) | 26 (81)
Pain - Abdomen (General disorders) | 5 (8) | 10 (16)
Dysuria (Renal and urinary disorders) | 4 (4) | 5 (5)
Pain - Back (General disorders) | 4 (9) | 0 (0)
Pain - Chest (General disorders) | 2 (2) | 0 (0)
Pain - Head (General disorders) | 2 (4) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 8 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (17)
Pain - Rectum (General disorders) | 3 (3) | 4 (5)
Platelets (Blood and lymphatic system disorders) | 10 (27) | 13 (31)
Proctitis (Gastrointestinal disorders) | 2 (2) | 3 (4)
Proteinuria (Renal and urinary disorders) | 8 (29) | 9 (17)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 8 (18) | 10 (12)
Neuropathy - Sensory (Nervous system disorders) | 18 (58) | 18 (65)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5)
Taste Alteration (Gastrointestinal disorders) | 6 (13) | 4 (12)
Ulceration (Skin and subcutaneous tissue disorders) | 7 (10) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 3 (4) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (10) | 10 (16)
Watery Eye (Eye disorders) | 3 (7) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 7 (19) | 5 (12)
Wound Complication (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.